CLINICAL TRIAL: NCT06013553
Title: The Effect of Aerobic Exercise on Neutrophil-Lymphocyte Ratio, Platelet-Lymphocyte Ratio and Lymphocyte-Monocyte Ratio in Burn Patients: A Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Murat Ali ÇINAR, assistive professor, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAC2023
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Burns; Physiotherapy; Aerobic Exercises
Keywords: burns,; neutrophil lymphocyte ratio; Platelet-Lymphocyte ratio; Lymphocyte Monocyte ratio
MeSH Terms: conditions — Burns | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Standard physiotherapy (1st Group): It comprised of parameters such as early mobilization and ambulatory training, pulmonary physiotherapy, active and passive normal joint movement exercises.
  Interventions: Other: Control Group
- Experimental: Aerobic Exercises group (Experimental): Aerobic exercise will be given with bicycle ergometer in addition to Standard physiotherapy (It comprised of parameters such as early mobilization and ambulatory training, pulmonary physiotherapy, active and passive normal joint movement exercises)
  Interventions: Other: Aerobic Exercises group

INTERVENTIONS:
Other: Control Group — It comprised of parameters such as early mobilization and ambulatory training, pulmonary physiotherapy, active and passive normal joint movement exercises.
  Arms: control group
Other: Aerobic Exercises group — Standard physiotherapy + bicycle ergometer: In addition to the standard therapy, a bicycle ergometer for 20 minutes 5 days a week will be given.
  Patients will turn the pedals of the bicycle while sitting on the edge of the bed.
  In this protocol, a portable bicycle with adjustable pedal system, which can be placed on the edge of the bed, will be used.
  "Ratings of perceived exertion (RPE)" will be used to determine the intensity of aerobic activity. According to the RPE, 10-12 strength exercises will be given
  Arms: Experimental: Aerobic Exercises group

SUMMARY:
In the study, it was planned to investigate the Effect on Neutrophil-Lymphocyte Ratio, Platelet-Lymphocyte Ratio and Lymphocyte-Monocyte Ratio in burn patients by creating 2 different exercise groups. The aim of this study is to investigate the effect of aerobic exercise on neutrophil-lymphocyte ratio, platelet-lymphocyte ratio and lymphocyte-monocyte ratios in burn patients.

DETAILED DESCRIPTION:
Burn injuries are a trauma that is seen due to causes such as flame, hot liquid, radiation, chemical, cold or electricity and causes destruction in the skin and/or organic tissues due to energy transfer.

Burn injuries cause profound hypermetabolic and catabolic responses that can last for months or even years. Especially in burn patients with involvement of more than 20% of the total body surface area (TVSA), lipolysis, proteolysis, glycolysis, and hyperdynamic and high fever, Many severe hypermetabolic responses are seen. These hypermetabolic responses seen in patients lead to decrease in lean muscle mass, inflammation, deterioration of cardiovascular, endocrine and glucose systems, coagulopathy, deterioration of fibrinolytic activity, decrease in functional capacity, delay in wound healing, weakening of the immune system and serious mortality.

In severely burned patients, the resting metabolic rate may exceed 140% of normal.

Various parameters are used to monitor all these systemic responses of the burn. Various scores have been developed in the clinic, especially using inflammatory cells such as neutrophils, monocytes, lymphocytes and platelets. In the literature, major diseases such as cancer, heart diseases and burns It has been stated that a systemic inflammation occurs due to trauma and calculations of neutrophil-lymphocyte ratio, platelet-lymphocyte ratio and lymphocyte-monocyte ratios are prognostic indicators.

Exercise in burn patients; It is a highly effective method with high evidence value in minimizing the effects of the hypermetabolic response caused by the burn, preventing muscle atrophy, increasing the pulmonary function and functional capacity, reducing the inflammatory response and healing the burn.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

Conscious patients Enterally fed >18 years old

Exclusion Criteria:

With inhalation burn In addition to existing burn trauma, those with other trauma (fracture, loss of limb, etc.) Organ dysfunctions or multiple organ failure History of chronic diseases such as diabetes, cholesterol and blood pressure

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Neutrophil lymphocyte ratio | Each participant will be evaluated for 6 weeks
  blood test
Platelet-Lymphocyte ratio | Each participant will be evaluated for 6 weeks
  blood test
Lymphocyte Monocyte ratio | Each participant will be evaluated for 6 weeks
  blood test

CONTACTS AND LOCATIONS:
Overall Officials: MURAT A ÇINAR, DR, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jeschke MG, van Baar ME, Choudhry MA, Chung KK, Gibran NS, Logsetty S. Burn injury. Nat Rev Dis Primers. 2020 Feb 13;6(1):11. doi: 10.1038/s41572-020-0145-5. PMID 32054846
- [Result] Romero SA, Moralez G, Jaffery MF, Huang M, Cramer MN, Romain N, Kouda K, Haller RG, Crandall CG. Progressive exercise training improves maximal aerobic capacity in individuals with well-healed burn injuries. Am J Physiol Regul Integr Comp Physiol. 2019 Oct 1;317(4):R563-R570. doi: 10.1152/ajpregu.00201.2019. Epub 2019 Aug 21. PMID 31433672
- [Result] Nielson CB, Duethman NC, Howard JM, Moncure M, Wood JG. Burns: Pathophysiology of Systemic Complications and Current Management. J Burn Care Res. 2017 Jan/Feb;38(1):e469-e481. doi: 10.1097/BCR.0000000000000355. PMID 27183443
- [Result] Cinar MA, Bayramlar K, Erkilic A, Gunes A, Yakut Y. The effects of early physiotherapy on biochemical parameters in major burn patients: A burn center's experience. Ulus Travma Acil Cerrahi Derg. 2019 Sep;25(5):461-466. doi: 10.5505/tjtes.2018.05950. PMID 31475319
- [Result] Flores O, Tyack Z, Stockton K, Paratz JD. The use of exercise in burns rehabilitation: A worldwide survey of practice. Burns. 2020 Mar;46(2):322-332. doi: 10.1016/j.burns.2019.02.016. Epub 2019 Dec 18. PMID 31864784
- [Derived] Cinar MA, Erkilic A. Effect of aerobic exercise on neutrophil-lymphocyte ratio, platelet-lymphocyte ratio, and lymphocyte-monocyte ratio in burn patients: A randomized controlled trial. J Plast Reconstr Aesthet Surg. 2024 Aug;95:199-206. doi: 10.1016/j.bjps.2024.05.032. Epub 2024 Jun 5. PMID 38936330